CLINICAL TRIAL: NCT02249377
Title: Clinical Outcomes of Platelet Rich Plasma Injection Versus Corticosteroid Injection for Baker's Cyst
Brief Title: PRP vs Corticosteroid in Baker's Cyst
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-00457
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Baker's Cyst
Keywords: Baker's Cyst
MeSH Terms: conditions — Popliteal Cyst | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelets-Rich-Plasma Group (Experimental): Patients will be asked to stop taking any type of anti-inflammatory medication from 7 days before the procedure to 2 weeks after and fasting for 3 hours before the procedure. At the moment of the procedure, the radiology team will draw 60ml of venous blood from the patient, the blood will be processed with different components of the PRP kit and centrifuged in the SmartPrep PRP machine, to obtain the PRP. The patient is then scanned prone using a linear 14 or 9 megahertz (MHz) transducer. A 20 Gauge spinal needle is usually employed for purposes of aspiration. Sterile saline will be used to confirm needle placement in the cyst in lieu of lidocaine and then inject the PRP by the radiologist.
  Interventions: Other: Platelets-Rich-Plasma
- Corticosteroid group: (Active Comparator): Patients will be asked to stop taking any kind of anti-inflammatory medication from 7 days before the procedure to 2 weeks after but fasting in this group won't be required. An ultrasound guided aspiration and triamcinolone (40 mg) diluted with lidocaine without epinephrine and ropivacaine will be used to anesthetize the tissues down to the cyst (including within the cyst for steroid injections). A compression bandage will be placed locally for 7 days. Investigators will monitor any side effect from the injection and treat the patients per standard care - this can include prescription of analgesics.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Other: Platelets-Rich-Plasma — Platelet-Rich Plasma
  Arms: Platelets-Rich-Plasma Group
Drug: Corticosteroid — Corticosteroid
  Arms: Corticosteroid group:

SUMMARY:
This is a Prospective study with Randomized patients into either Ultrasound-guided Platelets-Rich-Plasma injection and Ultrasound guided Corticosteroid Injection, with 3 months and 6 months follow ups after aspiration at our institution. There will be 25 patients in each group, including any patient with symptomatic baker's cyst.

DETAILED DESCRIPTION:
The treatment of Baker's Cysts are based on its presentation, asymptomatic cysts are currently managed conservatively, symptomatic cysts are treated with joint aspiration and Corticosteroid injection, which have shown according to literature a decrease of the cyst size in approximately two-thirds of patients within 2-7 days but only complete disappearance in approximately 7 %. Ultrasound guided cyst aspiration and Corticosteroid injection are also used with reduction of cyst's size with recurrence in 6 months of 19%. Surgical options to remove the cyst include, Open Resection with a recurrence of 50%, 25% of patients have motion limitation recurrence, 37% have wound healing problems or tense swelling of the calf and 75% of patients have joint pain lasting more than 2 days. Arthroscopic resection, with no recurrence in ultrasound performed 6 and 12 months after procedure, pain lasting more than 3 days in 28% of patients, mild hematoma in 7% of patients and 7% where converted into an open procedure

There is no study using ultrasound guided aspiration with platelet-rich-plasma injection (PRP). The rationale for the use of PRP is the belief that the additional platelets will exponentially increase the concentration and release of multiple growth and differentiation factors at the injury site to augment the natural healing process9. PRP does not have any described negative side effect due to the fact that is being prepared from subject's own blood, with no risk of allergy or cross infection, relatively easy for a practiced clinician, and reproducible.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old.
* Patients with baker's cyst who also present with at least one of the following: swelling, local pain or discomfort, limited range of motion or any other symptom directly caused by the baker's cyst.

Exclusion Criteria:

* Patients younger than 18 years old
* Local or Systemic active infection
* Active cancer treatment
* Immunodeficiency
* Diabetes
* Hypersensitivity or allergy to Corticosteroid or Lidocaine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Strauss, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Hospital for Joint Diseases - Center for Musculoskeletal Care, New York, New York, United States

REFERENCES:
- [Background] Handy JR. Popliteal cysts in adults: a review. Semin Arthritis Rheum. 2001 Oct;31(2):108-18. doi: 10.1053/sarh.2001.27659. PMID 11590580
- [Background] Johnson LL, van Dyk GE, Johnson CA, Bays BM, Gully SM. The popliteal bursa (Baker's cyst): an arthroscopic perspective and the epidemiology. Arthroscopy. 1997 Feb;13(1):66-72. doi: 10.1016/s0749-8063(97)90211-5. PMID 9043606
- [Background] Koroglu M, Callioglu M, Eris HN, Kayan M, Cetin M, Yener M, Gurses C, Erol B, Turkbey B, Parlak AE, Akhan O. Ultrasound guided percutaneous treatment and follow-up of Baker's cyst in knee osteoarthritis. Eur J Radiol. 2012 Nov;81(11):3466-71. doi: 10.1016/j.ejrad.2012.05.015. Epub 2012 Jun 20. PMID 22726355
- [Background] Ko S, Ahn J. Popliteal cystoscopic excisional debridement and removal of capsular fold of valvular mechanism of large recurrent popliteal cyst. Arthroscopy. 2004 Jan;20(1):37-44. doi: 10.1016/j.arthro.2003.10.017. PMID 14716277
- [Background] Acebes JC, Sanchez-Pernaute O, Diaz-Oca A, Herrero-Beaumont G. Ultrasonographic assessment of Baker's cysts after intra-articular corticosteroid injection in knee osteoarthritis. J Clin Ultrasound. 2006 Mar-Apr;34(3):113-7. doi: 10.1002/jcu.20210. PMID 16547992
- [Background] Omer Mei-Dan and Michael R. Carmont. Novel Applications of Platelet-Rich Plasma Technology in Musculoskeletal Medicine and Surgery. Oper Tech Orthop 22:56-63 © 2012 Elsevier
- [Background] Steven P. Arnoczky, Demetris Delos, Scott A. Rodeo. What Is Platelet-Rich Plasma? Oper Tech Sports Med 19:142-148 © 2011 Elsevier
- [Background] Mikel Sánchez, Javier Albillos, Francisco Angulo, Juanma Santisteban, Isabel Andia. Platelet-Rich Plasma in Muscle and Tendon Healing. Oper Tech Orthop 22:16-24 © 2012 Elsevier
- [Background] Andre F. Steinert, Kellie K. Middleton, Paulo H. Araujo, Freddie H. Fu. Platelet-Rich Plasma in Orthopaedic Surgery and Sports Medicine: Pearls, Pitfalls, and New Trends in Research. Oper Tech Orthop 22:91-103 © 2012 Elsevier
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] J.F. Kaux. Exuberant inflammatory reaction as a side effect of an infiltration of PRP. Médecine du sport (2) : tendinopathies (actualités) / Annals of Physical and Rehabilitation Medicine 56S (2013) e215-e221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
Started | 25 | 25
Completed | 0 | 1
Not Completed | 25 | 24

BASELINE CHARACTERISTICS:
Population: Study terminated due to lack of funding
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group: | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Outcome of Baker's Cysts With the Use of Platelets-Rich-Plasma Versus Corticosteroid
Description: Outcome measure will be determined through the use of the Visual Analogue Score (VAS) and the Rauschning and Lindgren criteria which are used to clinically evaluate the presence of the popliteal cysts, pain, posterior sense of tension in the popliteal fossa and its clinical importance for range of motion reduction. The Knee Injury and Osteoarthritis Outcome Score (KOOS) will be used to assess short and long term outcome of knee related conditions.
Time Frame: 6 Months
Population: The study was terminated due to lack of funding. Efforts were made to collect data, but were unsuccessful. No study data are available.
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Recurrence of Baker's Cysts Treated on Each Group
Description: as for outcome 1
Time Frame: 6 Months
Population: as for outcome 1
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Complications
Description: All disease signs and symptoms experienced by the patient, as defined as an Adverse Event (AE), Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE), and Unexpected Adverse Device Effect (UADE), will be recorded from questionnaires during each study visit.
Time Frame: 6 Months
Population: as for outcome 1
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Side Effects
Description: as for outcome 3
Time Frame: 6 Months
Population: as for outcome 1
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Study terminated due to lack of funding. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed as a result.
Arm/Group | Platelets-Rich-Plasma Group | Corticosteroid Group:
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT02249377/Prot_SAP_000.pdf